CLINICAL TRIAL: NCT06956339
Title: Evaluating Non-surgical Management of Acute Anterior Cruciate Ligament Rupture With a Novel BRACE Protocol Versus Early Surgical Reconstruction - a Comparative Effectiveness Randomised Controlled Trial
Brief Title: Cross Bracing Protocol Versus Surgery for Acute Anterior Cruciate Ligament Rupture
Acronym: EMBRACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMBRACE 31092
Record Dates: First submitted 2025-05-01; First posted 2025-05-04 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-04

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: anterior cruciate ligament; cross bracing; ACL healing; ACL; ACL reconstruction surgery
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The trial statisticians will remain blinded to treatment allocation until the Statistical Analysis Plan has been written, the database has been cleaned, a blinded data review has taken place and the database is ready for analysis.
  Radiologists grading follow-up MRIs will be blinded to participant details and group allocation, so they cannot discern people who were allocated to early surgery from those who had delayed surgery after being allocated to the bracing group. However, it is not possible to blind radiologists to the surgical status of participants (i.e. those who have undergone surgery vs those who have not) as surgical hardware is visible on MRI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery group (Active Comparator): Anterior cruciate ligament reconstruction surgery, undertaken within eight weeks of randomisation, and followed by 12 months of physiotherapist-supervised rehabilitation.
  Interventions: Procedure: Early anterior cruciate ligament surgery
- Bracing group (Experimental): A specialised bracing protocol to facilitate healing of the anterior cruciate ligament, including 4 weeks with the knee braced at 90 degrees, and 12 months of supervised physiotherapy rehabilitation.
  Interventions: Other: Novel bracing protocol

INTERVENTIONS:
Procedure: Early anterior cruciate ligament surgery — Participants randomised to early anterior cruciate ligament reconstruction surgery (ACLR) will be referred to a study orthopaedic surgeon. Participants will have surgery within 8 weeks of randomisation. The ACLR will reflect usual care for each surgeon. Participants will undergo routine preoperative care, including an anaesthetic consultation to assess fitness for surgery and general anaesthesia. Surgeons will choose their preferred surgical technique and graft, and treat concomitant injuries surgically if indicated and aligned with their usual practice. Participants will follow the surgeon's standard recommendations regarding post-operative care and appointments. Participants will be provided with 15 funded physiotherapy consultations within 12 months of surgery and undertake a physiotherapist-supervised goal-oriented exercise-based rehabilitation program.
  Arms: Surgery group
Other: Novel bracing protocol — Participants will undertake the Cross Bracing Protocol under the supervision of a study physiotherapist (23 funded physiotherapy sessions within 12 months). Medical oversight and venous thromboembolism prophylaxis will be provided by the study sports and exercise medicine physician.
  A specialised knee brace will be fitted within 21 days of ACL injury. The knee is kept at 90° flexion in the brace at all times for the first four weeks. The brace is then adjusted weekly by the physiotherapist to allow progressive increases in knee range (60-90° flexion at 5 weeks, 45-90° flexion at 6 weeks, 30° to full flexion at 7 weeks, 20° to full flexion at 8 weeks, 10° to full flexion at 9 weeks, unrestricted range at 10 weeks, brace off at 12 weeks). Whilst braced and after brace removal, the participant will undertake physiotherapist-supervised goal-oriented exercise-based rehabilitation within the available knee range.
  Arms: Bracing group

SUMMARY:
The aim of the EMBRACE clinical trial is to compare outcomes (knee pain, symptoms, function and quality of life) between people with anterior cruciate ligament (ACL) rupture who are managed with either a novel bracing protocol (Cross Bracing Protocol), or with ACL reconstruction surgery. The main question that the trial aims to answer is:

In individuals with acute ACL rupture, is management with the Cross Bracing Protocol more clinically effective and cost effective compared to early ACL reconstruction surgery?

180 people across five Australian cities, with a recent ACL injury, will be randomly allocated to one of two treatments.

1. Cross Bracing Protocol

   People who are allocated to the bracing treatment will:
   * wear a knee brace for 12 weeks
   * see a sports doctor
   * have 23 visits to a physiotherapist who will supervise their knee rehab over 12 months.
   * have two knee scans; 3 and 18 months after they enrol
2. Anterior Cruciate Ligament Reconstruction Surgery

People who are allocated to the surgery group will:

* have surgery within 8 weeks of enrolling in the study
* have 15 visits to a physiotherapist for their knee rehab over 12 months after surgery.
* have one knee scan 18 months after they enrol.

All participants will:

* complete surveys at the beginning and 3, 6, 12 and 18 months later so the main trial outcomes can be collected, as well as additional information about their knee.
* have knee imaging (Magnetic Resonance Imaging or MRI scan) so the overall condition of their knee can be assessed, as well as whether their ACL has healed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 to 40 years;
* Have a primary and acute ACL rupture (complete tear) confirmed by MRI scan;
* At least moderately active before the ACL injury (a score of 5 to 10 on the Tegner Activity Scale before the injury);
* Willing and able to give informed consent and participate fully in the interventions and assessment procedures;
* Willing and able to cover the out-of-pocket costs associated with ACLR surgery.

Exclusion Criteria:

* Have not completed the baseline questionnaire within 16 days of their initial ACL injury;
* Inability to read and speak English
* Concomitant knee injury diagnosed on MRI that requires surgical opinion and/or alterative treatment:

  i) Loose body ii) Unstable osteochondral defect iii) Intra-articular fracture that extends into the articular surface and requires reduction iv) Displaced and/or unstable meniscal tear v) Grade 2 and 3 posterolateral corner injury vi) High-grade medial collateral ligament (MCL) injury that requires treatment with a knee brace and/or surgery vii) Posterior cruciate ligament (PCL) injury (partial discontinuity with some preserved fibers or complete disruption)
* Severe disruption of ACL tissue visible on MRI:

  i) Gap distance ≥8mm and ≥ 25% of tissue displaced outside of intercondylar notch ii) Gap distance ≥8mm and ≥ 25% of femoral footprint avulsed iii) ≥ 25% of femoral footprint avulsed and ≥ 25% of tissue displaced outside of intercondylar notch iv) Complete femoral or tibial avulsion
* Concomitant patellofemoral joint dislocation diagnosed on MRI and/or self-reported history of recurrent patellofemoral joint instability or ≥1 patellofemoral joint dislocation;
* Self-reported episode of instability (i.e. 'giving way') since initial MRI that resulted in increased pain, swelling and reduced function (without a subsequent MRI to re-determine eligibility);
* Open growth plate of the femur and/or tibia visible on MRI;
* Past history of ACL injury on the ACL-injured knee;
* Past history of any surgery on ACL-injured knee;
* Breastfeeding, pregnancy or planned pregnancy within the first 12 weeks of the trial;
* Health conditions/medications that are contraindications for ACLR, CBP and/or use of anticoagulant (rivaroxaban) medication:

  i) Current deep vein thrombosis (DVT); ii) Past history of DVT and/or pulmonary embolism; iii) Diagnosed hypercoagulable disease (e.g., Protein C and Protein S deficiency, Factor 5 Leiden); iv) Significant renal/hepatic impairment (creatinine clearance <15mL/min, Child-Pugh score 10-15 (Class C)); v) Restless Legs Syndrome; vi) Current use of contraindicated medication (such as other anticoagulants, antiviral or oral anti-fungal medications); vii) Clinically significant active and/or recent bleeding (e.g., gastrointestinal, intracranial or haematuria); viii) At increased risk of clinically significant bleeding (e.g., significant inherited bleeding disorders, uncontrolled high blood pressure); ix) Other conditions requiring significant medical monitoring while anticoagulated, such as rheumatoid arthritis, type I or type II diabetes, autoimmune diseases; x) Self-reported body mass index (BMI) ≥40kg/m2, except in competitive athletes (defined as a pre-injury Tegner Activity Scale score of 7-10 and/or undertakes strength training/weightlifting two or more times per week); xi) Any known cardiovascular disease (history of stroke, coronary vascular disease); xii) Chronic obstructive pulmonary disease and/or chronic respiratory disease, except for controlled asthma; xiii) Acute infection of the knee or affected limb; xiv) Inflammatory arthropathy/arthritis; xv) knee osteoarthritis in the ACL-injured knee (assessed on acute knee MRI, defined as focal partial thickness cartilage loss or greater (at least ACLOAS grade 2 cartilage lesion2626) plus one or more definite osteophyte (at least ACLOAS grade 2 osteophyte26 xvi) Concurrent immunosuppressive illness (e.g., AIDS, cancer) and/or immunosuppressant usage; xvii) Connective tissue disorders (such as Ehlers-Danlos syndrome); xviii) Current systemic steroid usage; xix) Intravenous drug users and/or substance addiction.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Knee pain, symptoms, sport and recreational function, and knee-related quality of life as assessed by the Knee injury and Osteoarthritis Outcome Score (KOOS4) self-reported questionnaire. | Baseline and 6-, 12- and 18-months after randomisation
  An average of the four subscale scores is used for the overall KOOS4 score, from 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Anterior cruciate ligament-related quality of life as assessed by the Anterior Cruciate Ligament Quality of Life Scale (ACLQOL) self-reported questionnaire | Baseline and 6-, 12- and 18-months after randomisation
  Overall score ranges from 0 (worst) to 100 (best).
Return to pre-injury level of sport or activity as measured by the Tegner Activity Scale self-reported questionnaire | 6, 12 and 18 months after randomisation
  The Tegner Activity Scale is a self-reported single item questionnaire scored on an 11-item scale (0 (lower activity) -10 (higher activity). The number and proportion of participants who have returned to their same or higher level of sport or activity will be reported.
The number and proportion of participants satisfied with their knee function, where satisfaction with current knee function is assessed using a single item question | 6, 12 and 18 months after randomisation
Knee pain assessed using the Knee injury and Osteoarthritis Outcome Score (KOOS) Pain Subscale, with a score range from 0 (worst) to 100 (best). | Baseline and 6-, 12- and 18-months after randomisation
Knee symptoms assessed using the Knee injury and Osteoarthritis Outcome Score (KOOS) Symptoms Subscale, with a score range from 0 (worst) to 100 (best). | Baseline and 6-, 12- and 18-months after randomisation
Knee-related sport and recreational function assessed using the Knee injury and Osteoarthritis Outcome Score (KOOS) Sports and Recreational Activities Subscale, with a score range from 0 (worst) to 100 (best). | Baseline and 6-, 12- and 18-months after randomisation
Knee-related quality of life assessed using the Knee injury and Osteoarthritis Outcome Score (KOOS) Quality of Life Subscale, with a score range from 0 (worst) to 100 (best). | Baseline and 6-, 12- and 18-months after randomisation
Number of participants reporting with least one related serious adverse event during their 18-month period in the trial | From randomisation until the collection of the final data at 18 months
Number and proportion of participants reporting one or more anterior cruciate ligament re-rupture or graft rupture confirmed by MRI or arthroscopy | From randomisation until the collection of the final self-reported data at 18 months
Knee instability assessed by self-report of episodes of giving way of the anterior cruciate ligament injured knee | From randomisation until the collection of final data at 18 months
Fear of reinjury assessed using self-report of item 31 from the Anterior Cruciate Ligament Quality of Life Scale, ranging from 0 (extremely fearful) to 100 (no fear at all). | Baseline and 6-, 12- and 18-months after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Filbay, Principal Investigator — University of Melbourne
Locations (1):
- The University of Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
We will share all deidentified data that support published results of the trial. Additional data that have not been published will be withheld until at least six months after publication. Data will be made available as required for specific, approved analyses, where these comply with our ethical requirements and the planned secondary analysis is of sufficient methodological rigour. Data will be provided from locked, cleaned, and de- identified study database. Requests will be reviewed by the Principal Investigator prior to approval.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Once the paper has been published and subject to signing of a legal agreement and within the timeframe of the data retention period specified by the Human Research Ethics Committee.
Access Criteria: The investigators endorse the concept of data sharing to advance medical science. All requests for data sharing will be reviewed by the Principal Investigator to ensure no conflict with any planned sub analyses, that the planned secondary analysis is of sufficient methodological rigour, and to ensure that the data are shared in an ethical and protected manner. Data will be made available after review and approval by the Principal Investigator. Before any analysis, a signed Confidentiality Agreement and/or Data Sharing Agreement is required. Analyses that aim to improve management of anterior cruciate ligament injury for non-commercial purposes are eligible.
URL: https://healthsciences.unimelb.edu.au/departments/physiotherapy/chesm/projects/embrace